CLINICAL TRIAL: NCT05505422
Title: Randomized Trial of Routine Versus Selective Use of Intraoperative Extracorporeal Mechanical Support During Lung Transplantation : a Pilot Study
Brief Title: Routine Versus Selective Intraoperative ECMO in Lung Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-10663
Record Dates: First submitted 2022-08-09; First posted 2022-08-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Lung Transplant; Complications; Extracorporeal Circulation; Complications; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On demand ECMO (study group) (Experimental)
  Interventions: Device: On demand ECMO
- Routine ECMO (control group) (Active Comparator)
  Interventions: Device: Routine ECMO

INTERVENTIONS:
Device: Routine ECMO — Routine ECMO during lung tansplant
  Arms: Routine ECMO (control group)
Device: On demand ECMO — Selective, indication-based intraoperative cardiopulmonary support. In this group, the transplant will be planned without cardiopulmonary support. intraoperative ECMO will be used selectively based on hemodynamic and/or gas exchange abnormalities :
  1. Inability to maintain adequate hemodynamics and stable perfusion or oxygenation during surgery
  2. Prolonged high dose pressor required to maintain adequate perfusion
  3. A sustained drop in cerebral saturation > 25% of baseline despite initial attempts at optimization
  4. Inability to tolerate pulmonary artery clamping
  5. Inadequate gas exchange despite attempts at the optimization of ventilator parameters and treatments related to respiratory mechanics and ventilation/perfusion matching
  6. Inadequate exposure to the surgical field
  Arms: On demand ECMO (study group)

SUMMARY:
Intraoperative hemodynamic management is vital in the success of lung transplantation. Significant intraoperative hemodynamic compromise and hypoxic episodes may contribute to an increase in severe postoperative complications related to hypoperfusion, including cerebrovascular accidents, acute kidney injury, and mesenteric ischemia. In certain lung transplant recipients, intraoperative cardiopulmonary support is mandatory because certain factors would make "off-pump" transplants unsafe. These include severe pulmonary hypertension or severe ventricular dysfunction. In such patients, routine intraoperative support should be employed. However, it is possible to conduct the lung transplant without cardiopulmonary support in the remainder of patients who do not have severe pulmonary hypertension or right heart dysfunction. In such patients, the lung transplant may be started without cardiopulmonary support. However, cardiopulmonary support may be initiated "on-demand" if there is development or impending hemodynamic embarrassment or hypoxia. Conversely, the opposite approach would be to routinely conduct all lung transplant operations using cardiopulmonary support, which may also lead to specific ECMO-related complications.

The investigators question whether on demand intraoperative ECMO in patients with significant risk factors will produce severe postoperative complications in a rate similar to routine ECMO.

DETAILED DESCRIPTION:
Hypothesis: In patients where cardiopulmonary bypass (CPB) / ECMO is not mandatory, on-demand use of intra-operative ECMO is equivalent to routine use for patients undergoing lung transplant.

The study will be a prospective, randomized controlled trial. The investigators seek to compare outcomes of two different strategies of cardiopulmonary support during lung transplantation; routine support with ECMO versus selective (on-demand), indication- based support with ECMO. The allocation ratio will be 1:1. A multi-center trial is necessary to allow for a sufficient sample size. However, the investigators believe a pilot study is essential to determine feasibility before embarking on such a significant undertaking.

In this preliminary pilot study, recruitment will be limited to lung transplant patients at the Centre hospitalier de l'Universite de Montreal (CHUM). The primary purpose of the pilot study will be to define recruitment ability and assess the feasibility of conducting the study. Depending on the results of this pilot study, the next step would be to expand the study to multiple lung transplant centers to achieve an adequate sample size and power, allowing the investigators to answer the question of interest.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing lung transplant surgery during the study period (6 months)

Exclusion Criteria:

1. Inability to provide consent for the study or patient refusal
2. Retransplantation
3. Multi-organ transplantation
4. Lung transplant recipients where intraoperative support is mandatory and "off- pump" transplant would be unsafe:

   a. Severe pulmonary hypertension (PH):

   i. Systolic pulmonary artery pressure (PAP) ≥ 80 mm Hg on echocardiography, right heart catheterization, or pulmonary artery catheter measurement

   ii. Mean PAP ≥ 55 mm Hg on echocardiography, right heart catheterization, or pulmonary artery catheter measurement

   iii. The ratio of mean pulmonary to systemic artery pressure of more than 0.66

   b. Moderate to severe right ventricular (RV) hypokinesis or dysfunction

   c. Left ventricular dysfunction: Defined as ejection fraction (LVEF) < 50% on echocardiography, ventriculography, computed tomography (CT), or magnetic resonance imaging (MRI)

   d. Significant coronary artery disease (CAD)requiring stenting or surgical grafting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Study recruitment rate | 6 months after the onset of study

SECONDARY OUTCOMES:
Percentage of patients loss to follow-up | 1 year
The composite incidence of death, disabling stroke, grade 2 or 3 primary graft dysfunction at 72 hours, major bleeding (BARC grade 3a, 3b or 5), vascular complications, or stage II or III acute kidney injury at 14 days. | 14 days
Incidence of all-cause mortality at 30 days, 90 days, and one year | 1 year
Incidence of postoperative stroke / cerebrovascular accident | 14 days
Incidence of an Early major postoperative neurologic complication (EMPNC): This includes stroke, severe encephalopathy, and severe seizures diagnosed within 14 days after surgery. | 14 days
Incidence of severe postoperative complications. This is defined as Clavien-Dindo grade III complication or greater | 14 days

OTHER OUTCOMES:
Incidence and grade of primary graft dysfunction (PGD) at 0, 24, 48, and 72 hours | From the end of surgery up to 72 hours after surgery
Incidence of postoperative bleeding complications. The definition of bleeding complication is based on Bleeding Academic Research Consortium (BARC) classification | 14 days after surgery
Intraoperative blood product transfusion requirements | From the beginning of surgery to transfer to the intensive care unit
Perioperative blood product transfusion requirements | 14 days
  From the beginning of surgery to 14 days after surgery, including return to the operating room for subsequent surgeries
Intensive care unit and hospital length of stay in days | Beginning from the arrival to the intensive care unit immediately after surgery
Duration of mechanical ventilation in hours | Beginning from the arrival to the intensive care unit immediately after surgery, up to about 30 days
  BiPAP and CPAP are not considered mechanical ventilation. Tracheostomy is not considered mechanical ventilation if a ventilator is not needed.
Incidence of re-intubation | 14 days
Incidence of postoperative tracheostomy | 21 days
Incidence of acute kidney injury (AKI) within 14 days. The definition of AKI is based on Kidney Disease; improving global outcomes (KDIGO) classification | 14 days
Incidence of vascular complications | 14 days
Forced expiratory volume at 1 second (FEV1) at 1 year | 1 year
Incidence of stroke | 1 year
Incidence of acute rejection episodes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Basil Nasir, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasir BS, Weatherald J, Ramsay T, Cypel M, Donahoe L, Durkin C, Schisler T, Nagendran J, Liberman M, Landry C, Overbeek C, Moore A, Ferraro P. Randomized trial of routine versus on-demand intraoperative extracorporeal membrane oxygenation in lung transplantation: A feasibility study. J Heart Lung Transplant. 2024 Jun;43(6):1005-1009. doi: 10.1016/j.healun.2024.02.1454. Epub 2024 Feb 28. PMID 38423414